CLINICAL TRIAL: NCT02538952
Title: Evaluating Performance, Impact, and Operational Challenges of GeneXpert Use for TB Case Finding Among HIV-infected Persons in Botswana During 2012-2013: The Xpert Package Rollout Evaluation Study (XPRES)
Brief Title: Evaluating Accuracy, Impact, and Operational Challenges of GeneXpert Use for TB Case Finding Among HIV-infected Persons
Acronym: XPRES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Botswana Ministry of Health (Other Government); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CDC-CGH-6294
Record Dates: First submitted 2015-08-20; First posted 2015-09-02 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2017-07

CONDITIONS: Tuberculosis; Human Immunodeficiency Virus
Keywords: GeneXpert; Tuberculosis; Human immunodeficiency virus; Diagnostic accuracy; Impact
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome; Tooth, Impacted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Xpert package (Experimental): There are three phases to this stepped-wedge trial: (1) the retrospective cohort (standard of care) phase, (2) the active comparator phase, where intensified TB case finding (ICF) interventions are in place but no Xpert device, and (3) the "experimental phase" of full Xpert package implementation that includes both ICF interventions and Xpert device activation. Interventions in the experimental phase therefore include: (a) adoption of the WHO-recommended 4-symptom TB screen for adults; (b) situating trained TB case-finding nurses in the 22 facilities; (c) training health facility personnel in TB diagnostic algorithms; and (d) Xpert device activation. The combination of the ICF interventions and rollout of the Xpert device is referred to as the "Xpert package" in this protocol.
  Interventions: Device: Xpert device; Other: Intensified TB Case Finding (ICF)
- Active comparator (Active Comparator): There are three phases to this stepped-wedge trial: (1) the retrospective cohort (standard of care) phase, (2) the active comparator phase, where intensified TB case finding (ICF) interventions are in place but no Xpert device, and (3) the "experimental phase" of full Xpert package implementation that includes both ICF interventions and Xpert device activation. Interventions in the active comparator phase therefore include only: (a) adoption of the WHO-recommended 4-symptom TB screen for adults; (b) situating trained TB case-finding nurses in the 22 facilities; and (c) training health facility personnel in TB diagnostic algorithms. There is no Xpert device activation in this phase. Only standard of care microscopy-based TB diagnostic algorithms are available during this phase.
  Interventions: Other: Intensified TB Case Finding (ICF)
- Standard of Care (No Intervention): There are three phases to this stepped-wedge trial: (1) the retrospective cohort (standard of care) phase, (2) the active comparator phase, where intensified TB case finding (ICF) interventions are in place but no Xpert device, and (3) the "experimental phase" of full Xpert package implementation that includes both ICF interventions and Xpert device activation. There are no interventions in the standard of care arm (retrospective cohort). There are no ICF interventions and no Xpert device activations in this phase. Only the standard of care TB case finding procedures and microscopy-based TB diagnostic algorithm are available during this phase.

INTERVENTIONS:
Device: Xpert device — Interventions in the "Experimental phase" of this stepped-wedge trial include: (a) ensuring WHO-recommended TB screening adopted, (b) situating trained TB case finding nurses in the clinics, (c) training clinic personnel in the TB diagnostic algorithms, and (d) activation of the Xpert diagnostic device.
  Arms: Xpert package
Other: Intensified TB Case Finding (ICF) — Interventions in the active comparator phase of this stepped wedge trial only include: (a) adoption of the WHO-recommended 4-symptom TB screen for adults; (b) situating trained TB case-finding nurses in the 22 facilities; and (c) training health facility personnel in TB diagnostic algorithms. There is no Xpert device activation in this phase. Only the standard of care microscopy algorithm (smear microscopy and chest x-ray) are available during this phase.
  Arms: Active comparator; Xpert package

SUMMARY:
Background: In Botswana, as in the rest of sub-Saharan Africa, undiagnosed TB or TB diagnosed late in the course of disease is thought to be the most common cause of death among HIV-infected persons.

Interventions for Evaluation: The Xpert MTB/RIF assay for the GeneXpert platform (Xpert) has a TB diagnostic sensitivity of 82.4%, significantly superior to that of smear microscopy (44.6%). In line with WHO guidelines, the Botswana Ministry of Health (MOH) and CDC rapidly rolled out the Xpert device and a new Xpert-based diagnostic algorithm in service of 22 HIV care and treatment clinics. To maximize impact of the Xpert device in improving detection of active TB, Xpert rollout was preceded by strengthening of TB screening procedures by: (1) adopting the WHO-recommended 4-symptom TB screen for adults; (2) situating trained TB case-finding nurses in facilities; and (3) training health facility personnel in TB diagnostic algorithms. The combination of these strengthened TB screening procedures and rollout of the Xpert device is referred to as the "Xpert package" in this protocol.

Key Evaluation Objectives: The protocol has two key objectives: (1) to evaluate whether the new MOH-recommended Xpert-based TB diagnostic algorithm for new adult HIV clinic enrollees is more sensitive than the pre-Xpert smear-microscopy-based algorithm in diagnosing culture-positive TB disease; and (2) to evaluate the impact of the whole "Xpert package" on all-cause mortality during the first 6 months of ART, among adult patients.

Design: Stepped-wedge cluster randomized trial. Sample Size: 6,136 patients were prospectively enrolled to meet the first primary objective. A retrospective cohort of 10,131 persons was also enrolled to meet the second objective. Projected power to meet both objectives is >80%.

Time line: Prospective cohort enrollment started in July 2012 and was complete by March 2014. Retrospective cohort enrollment was complete by March 2015. Patient follow-up and data entry will be complete in March 2016 at which time analysis to answer the first two primary study questions will be possible.

DETAILED DESCRIPTION:
Background: In Botswana, as in the rest of sub-Saharan Africa, undiagnosed tuberculosis (TB) or TB diagnosed late in the course of disease is thought to be the most common cause of death among HIV-infected persons receiving antiretroviral therapy (ART) as well as those not yet on ART. Common reasons for failure to diagnose TB early, include: (1) failure to appropriately screen HIV-infected patients for TB; and (2) difficulty in diagnosing TB with traditional diagnostic methods.

Public Health Intervention: The recent development of the Xpert MTB/RIF assay for the GeneXpert platform (Xpert) has revolutionized TB diagnostic capability for clinicians managing HIV-infected patients. Among HIV-infected adults, TB diagnostic sensitivity of Xpert (82.4%) has been proven superior to that of smear microscopy (44.6%). In line with World Health organization (WHO) guidelines, the Botswana Ministry of Health (MOH) and the United States Centers for Disease Control and Prevention (CDC), initiated a project in July 2012 to rapidly rollout 13 Xpert devices in service of 22 HIV care and treatment clinics while simultaneously initiating an evaluation to answer important operational research questions that can inform future national scale-up. To maximize the impact of the Xpert device in improving detection of active TB, the Xpert rollout was preceded by strengthening of TB screening procedures by: (1) ensuring the 22 HIV care and treatment clinics adopted the WHO-recommended four-symptom TB screen for adults; (2) situating trained TB case-finding nurses in all 22 facilities; and (3) training health facility personnel in both smear-microscopy-based and Xpert-based TB diagnostic algorithms. The combination of these strengthened TB screening procedures and rollout of the Xpert device is referred to as the "Xpert package" in this proposal.

Key Evaluation Objectives: The evaluation component of this project has two key objectives: (1) to evaluate whether the new MOH-recommended Xpert-based pulmonary TB diagnostic algorithm (including Xpert testing of sputum samples for all TB suspects and chest x-ray for Xpert-negative TB suspects) is more sensitive than the pre-Xpert smear-microscopy-based algorithm (smear microscopy and chest x-ray for smear-negative TB suspects) in diagnosing culture-positive TB disease; and (2) to evaluate the impact of the whole "Xpert package" on all-cause mortality during the first six months of ART, among adult patients.

Rationale for the First Evaluation Objective: Although it is expected that the Xpert-based TB diagnostic algorithm will be both more sensitive and more specific than the pre-Xpert algorithm, superiority of the Xpert- over the microscopy-based algorithm in Botswana has not yet been evaluated.

Rationale for the Second Evaluation Objective: In Botswana, undiagnosed TB or TB diagnosed late in the course of disease is thought to be the most common cause of death among HIV-infected persons receiving antiretroviral therapy (ART). The Xpert package could conceivably reduce TB-related mortality by ensuring all patients are screened for TB and ensuring TB suspects have access to a sensitive TB test (Xpert). Since the start of our Botswana stepped wedge trial in 2012, two separate but related randomized trials in Africa, the TB-NEAT study and the XTEND trial, have fallen short of demonstrating an association between use of Xpert for patients with symptoms of TB and reduced TB mortality. However, limitations in both these trials mean that the question of whether Xpert can reduce early ART mortality has not been definitively answered.

Design: Because the Xpert package is expected to have a beneficial effect for patients enrolling in the 22 study clinics, a phased rollout of the Xpert device using a stepped wedge design was chosen. Prior to Xpert device rollout, all 22 facilities initiated the intensified TB screening procedures simultaneously. Subsequently, 13 Xpert devices were activated in a step-wise manner over nine months with either one or two Xpert devices activated per month and the order of Xpert device rollout randomly assigned.

This step-wedge design involved enrollment of three cohorts:

1. Prospective cohort A (enrolled pre-Xpert device rollout): All patients who attended one of the 22 HIV clinics for the first time after study start (July 31, 2012), but before Xpert device rollout, were eligible for this cohort.
2. Prospective cohort B (enrolled post-Xpert device rollout): All patients who attend one of the 22 HIV clinics for the first time after Xpert device rollout were eligible for this cohort.
3. Retrospective cohort: All patients who initiated ART at one of the 22 HIV clinics for the first time in the 24 months before study start.

To answer the first primary study question, sensitivity of the pre- Xpert TB diagnostic algorithm in prospective cohort A will be compared with the post- Xpert algorithm sensitivity in prospective cohort B.

To answer the second primary study question, the investigators will compare 6-month ART mortality rates of ART enrollees in the retrospective cohort with 6-month ART mortality rates in prospective cohort B.

Power to Answer First Primary Study Question: Fisher's Exact Test sample size formula for comparing two proportions and Proc Power features in SAS version 9.2. software, were used to estimate study power. Power estimates were adjusted for the expected design effect to account for intra-cluster correlation. For design effect calculations, an intra-class correlation of 0.05 was assumed. With an anticipated sample size of 6,136 prospective enrollees (1,878 pre-Xpert and 4,258 post-Xpert), the study is estimated to have >80% power to detect pre- versus post-Xpert TB diagnostic sensitivities, assuming a culture-positive TB prevalence of 4% among prospective cohort enrollees, if pre-Xpert sensitivity is ≤52.5% and post-Xpert sensitivity is ≥82.5%.

Power to Answer Second Primary Study Question: As of August 2015, 10,131 ART patient medical records had been abstracted for the retrospective cohort. Published literature suggests pre-Xpert 6-month ART mortality rates should be about 15 per 100 person years (PY). Using published cluster randomized trial (CRT) power formulae adapted for stepped wedge trials and anticipated study sample sizes, the study has >80% power to detect a difference in 6-month all-cause ART mortality between cohorts R and B of 50% if cohort R mortality is ≥6/100 PY and of 40% if cohort R mortality is ≥13/100 PY.

Procedures: All 22 health facilities were assessed prior to training to troubleshoot potential logistical barriers to successful study implementation. All personnel involved in study procedures were trained before study start and closely supervised during implementation. Patients enrolled in the prospective cohorts are being followed for six months after HIV clinic enrollment, or through the end of TB treatment, whichever is later. Tracing of ART patients in retrospective and prospective cohorts, who are documented as late for appointments or lost to follow-up (missed last scheduled appointment by >60 days) has been performed according to national guidelines to facilitate estimation of true 6-month ART mortality.

Time line: Prospective cohort enrollment started in July 2012 and was complete by March 2014. Retrospective cohort enrollment was complete by March 2015. Patient follow-up and data entry will be complete in March 2016 at which time analysis to answer the first two primary study questions will be possible.

ELIGIBILITY:
Prospective cohorts:

Inclusion Criteria:

* All new HIV clinic enrollees who meet consent requirements.

Exclusion Criteria:

* Prisoners

Retrospective cohort:

Inclusion Criteria:

* All patients starting antiretroviral therapy at a study clinic in the 24 months before study start.

Exclusion Criteria:

* Prisoners

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18696 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
TB diagnostic sensitivity among adults (>12 years old). Sensitivity proportions will be estimated using laboratory data on TB diagnoses (see "Description" below). | Patients will be followed for an average of about 6 months each, and TB diagnostic sensitivity will be estimated at each clinical visit where the patient tests culture-positive for TB, with clinic visits occuring every one to 3 months.
  TB diagnostic algorithm sensitivity will be estimated in the pre-Xpert and post-Xpert time periods of this stepped wedge design, among adults (>12 years old). Sensitivity is the proportion of culture-positive TB cases correctly diagnosed with TB using the relevant diagnostic algorithm. The denominator is all culture-confirmed TB cases and the numerator the number of culture-confirmed TB cases that were correctly identified as positive by the relevant TB diagnostic algorithm.
All-cause mortality | Patients will be followed for an average of about 6 months each, with vital status assessed across the 6 month follow-up period.
  All-cause 6-month mortality among adult antiretroviral therapy enrollees will be compared between the pre-Xpert retrospective cohort and the post-Xpert package cohorts.

SECONDARY OUTCOMES:
Clinician TB screening compliance. Compliance proportions will be estimated using data from study questionnaires (see "Description" below). | Patients will be followed for an average of about 6 months each, with clinician TB screening compliance assessed at each clinic visit, which should occur every one to 3 months.
  Clinician TB screening compliance will be compared between the pre-Xpert and post-Xpert cohorts. This is the proportion of clinic visits that the TB screening algorithm for adults was correctly administered by the attending clinician. The denominator is the number of clinic visits and the numerator is the number of occasions that the TB screening algorithm was completely and correctly administered.
The proportion of patients screening positive for TB at the HIV clinic enrollment visit. Proportions screening positive will be estimated using data from study questionnaires (see "Description" below). | Patients will be followed for an average of about 6 months each, and the proportion screening positive for TB will be estimated at each clinical visit, including the first clinic visit, with clinic visits occuring every one to 3 months.
  The proportion of HIV clinic enrollees, who screen positive for TB, will be compared between the pre-Xpert and post-Xpert cohorts. The denominator of the proportion will be the number of patients screened for TB at the HIV clinic enrollment visit, and the numerator will be the number of patients screening positive for TB at the HIV clinic enrollment visit.
The proportion of patients diagnosed with TB at HIV clinic enrollment. Proportions diagnosed with TB will be estimated using data from study questionnaires and laboratory tests. | Patients will be followed for an average of about 6 months each, and the proportion diagnosed with TB will be estimated at each clinical visit, with clinic visits occuring every one to 3 months.
  The proportion of HIV clinic enrollees, who are diagnosed with TB following tests conducted at the enrollment visit, will be compared between the pre-Xpert and post-Xpert cohorts. The denominator will be the number of patients attending the HIV clinic enrollment visit, and the numerator will be the number of patients diagnosed with TB at the HIV clinic enrollment visit.
TB diagnostic sensitivity among children (<=12 years old). Sensitivity proportions will be estimated using laboratory data on TB diagnoses (see "Description" below). | Patients will be followed for an average of about 6 months each, and TB diagnostic sensitivity will be estimated at each clinical visit where the patient tests culture-positive for TB, with clinic visits occuring every one to 3 months.
  TB diagnostic algorithm sensitivity will be estimated in the pre-Xpert and post-Xpert time periods of this stepped wedge design, among children (<=12 years old). Sensitivity is the proportion of culture-positive TB cases among children correctly diagnosed with TB using the relevant diagnostic algorithm. The denominator is all culture-confirmed TB cases among children and the numerator the number of culture-confirmed TB cases that were correctly identified as positive by the relevant TB diagnostic algorithm.
TB screening algorithm sensitivity among children (<=12 years old). Sensitivity proportions will be estimated using laboratory data on TB diagnoses and questionnaire data on the screening algorithm (see "Description" below). | Patients will be followed for an average of about 6 months each, and TB diagnostic sensitivity will be estimated at each clinical visit where the patient tests culture-positive for TB, with clinic visits occuring every one to 3 months.
  MOH-recommended TB screening algorithm sensitivity will be estimated among children (<=12 years old). Sensitivity is the proportion of culture-positive TB cases correctly identified as potentially having TB using the MOH-recommended, 6-symptom, TB screening algorithm for children. The denominator is all culture-confirmed TB cases among children, and the numerator is the number of culture-confirmed TB cases that were correctly identified as potentially having TB by the 6-symptom, TB screening algorithm for children.
Diagnostic sensitivity of Xpert in diagnosing culture-positive drug resistant TB. | Patients will be followed for an average of about 6 months each, and TB diagnostic sensitivity will be estimated at each clinical visit where the patient tests culture-positive for drug resistant TB, with clinic visits occuring every one to 3 months.
  The study will estimate the sensitivity of the Xpert-based TB diagnostic algorithm in identifying drug resistant TB. The denominator is all culture-confirmed TB cases with genotypic or phenotypic drug resistance, and the numerator is the number of culture-confirmed drug resistant TB cases that were correctly identified as rifampicin resistant by the Xpert-based diagnostic algorithm.
TB incidence | Patients will be followed for an average of about 6 months each, and TB incidence will be estimated at each clinical visit, with clinic visits occuring every one to 3 months.
  TB incidence among adult antiretroviral therapy enrollees will be compared between the pre-Xpert cohorts and the post-Xpert package cohorts.
TB treatment outcomes. The incidence rate will be estimated using data from study questionnaires (see "Description" below). | Patients will be followed for an average of about 6 months each, and TB treatment outcomes will be estimated at each clinical visit, with clinic visits occuring every one to 3 months.
  TB treatment outcomes among HIV clinic enrollees will be compared between the pre-Xpert cohorts and the post-Xpert package cohorts. Possible treatment outcomes include "Cured", "Completed Treatment", "Died", "Treatment failure", "Defaulted/Lost-to-follow-up/missing", "Transferred out", and "Treatment ongoing".
Hospitalization rates. Incidence of hospitalization rates will be estimated from study questionnaires. | Patients will be followed for an average of about 6 months each, and the hospitalization outcome will be measured at each clinical visit, with clinic visits occuring every one to 3 months.
  Hospitalization rates among adult antiretroviral therapy enrollees in the first 6 months of ART will be compared between the pre-Xpert cohorts and the post-Xpert package cohorts.
Xpert diagnostic sensitivity. Sensitivity proportions will be estimated using laboratory data on TB diagnoses (see "Description" below). | Patients will be followed for an average of about 6 months each, and TB diagnostic sensitivity will be estimated at each clinical visit where the patient tests culture-positive for TB, with clinic visits occuring every one to 3 months.
  Variations in Xpert diagnostic accuracy by location (point of care versus lab-based), and over time, will be explored. Sensitivity is the proportion of culture-positive TB cases correctly diagnosed with TB using the relevant diagnostic algorithm. The denominator is all culture-confirmed TB cases and the numerator the number of culture-confirmed TB cases that were correctly identified as positive by the relevant TB diagnostic algorithm.
The proportion of attempts to use Xpert where Xpert was considered inoperable. These data will be obtained from study questionnaires. | Patients will be followed for an average of about 6 months each, and Xpert fuctionality be estimated at each clinical visit where the patient screens positive for TB and provides a sputum sample, with clinic visits occuring every one to 3 months.
  The study will estimate what proportion of attempts to use Xpert where Xpert was considered inoperable for any duration of time.
Median turnaround time for sputum samples from the time of sample collection to the time the patient was initiated on TB treatment. These data will be obtained from study questionnaires. | Patients will be followed for an average of about 6 months each, and turnaround times for sputum samples will be estimated at each clinical visit where the patient provides a sputum sample, with clinic visits occuring every one to 3 months.
  The median time from the time of sputum sample collection to the time of TB treatment initiation will be estimated using study questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Alyssa Finlay, MD, Principal Investigator — CDC Botswana; Tedd V Ellerbrock, MD, Principal Investigator — CDC Atlanta; Andrew F Auld, MBChB, MSc, Principal Investigator — CDC Atlanta; Tefera Agizew, MD, MPhil, Principal Investigator — CDC Botswana
Locations (1):
- 22 HIV care and Treatment clinics in Botswana, Multiple Locations, Multiple, Botswana

IPD SHARING:
Plan to Share IPD: Undecided
IRB-approved protocols and CDC regulations will be followed.

REFERENCES:
- [Derived] Auld AF, Fielding K, Agizew T, Maida A, Mathoma A, Boyd R, Date A, Pals SL, Bicego G, Liu Y, Shiraishi RW, Ehrenkranz P, Serumola C, Mathebula U, Alexander H, Charalambous S, Emerson C, Rankgoane-Pono G, Pono P, Finlay A, Shepherd JC, Holmes C, Ellerbrock TV, Grant AD. Risk scores for predicting early antiretroviral therapy mortality in sub-Saharan Africa to inform who needs intensification of care: a derivation and external validation cohort study. BMC Med. 2020 Nov 9;18(1):311. doi: 10.1186/s12916-020-01775-8. PMID 33161899
- [Derived] Auld AF, Agizew T, Mathoma A, Boyd R, Date A, Pals SL, Serumola C, Mathebula U, Alexander H, Ellerbrock TV, Rankgoane-Pono G, Pono P, Shepherd JC, Fielding K, Grant AD, Finlay A. Effect of tuberculosis screening and retention interventions on early antiretroviral therapy mortality in Botswana: a stepped-wedge cluster randomized trial. BMC Med. 2020 Feb 11;18(1):19. doi: 10.1186/s12916-019-1489-0. PMID 32041583
- [Derived] Agizew T, Chihota V, Nyirenda S, Tedla Z, Auld AF, Mathebula U, Mathoma A, Boyd R, Date A, Pals SL, Lekone P, Finlay A. Tuberculosis treatment outcomes among people living with HIV diagnosed using Xpert MTB/RIF versus sputum-smear microscopy in Botswana: a stepped-wedge cluster randomised trial. BMC Infect Dis. 2019 Dec 16;19(1):1058. doi: 10.1186/s12879-019-4697-5. PMID 31842773
- [Derived] Auld AF, Agizew T, Pals S, Finlay A, Ndwapi N, Boyd R, Alexander H, Mathoma A, Basotli J, Gwebe-Nyirenda S, Shepherd J, Ellerbrock TV, Date A. Implementation of a pragmatic, stepped-wedge cluster randomized trial to evaluate impact of Botswana's Xpert MTB/RIF diagnostic algorithm on TB diagnostic sensitivity and early antiretroviral therapy mortality. BMC Infect Dis. 2016 Oct 26;16(1):606. doi: 10.1186/s12879-016-1905-4. PMID 27782821
- See also: Trial findings reported at the Conference on Retroviruses and Opportunistic Infections (CROI) 2018. — http://www.croiconference.org/sessions/effect-tb-screening-and-retention-interventions-early-art-mortality-botswana